CLINICAL TRIAL: NCT06499584
Title: The Functional Role of Cochlear Synaptopathy for Speech Coding in the Brain
Brief Title: Study of the Fine Structure and Temporal Envelope of the Human Cochlea in Response to Human Vocalizations
Acronym: CosySpeech
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO23102
Record Dates: First submitted 2024-06-06; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Structure Cochlea; Temporal Envelope Cochlea
Keywords: Hearing Loss; Deafness; Micro vascular decompression; Otoneurosurgery; Retrosigmoid approach
MeSH Terms: conditions — Hearing Loss; Deafness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal hearing patients (Experimental): free of sensorineural hearing loss, defined by mean hearing thresholds of less than or equal to 20 dB HL in air conduction pure tone audiometry, bilaterally on the side of the operated ear and on the non-operated side at 0.5, 1, 2 and 4 kHz.
  Interventions: Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode
- hearing impaired patients (Experimental): with sensorineural hearing loss defined by average hearing thresholds between 21 dB HL and 40 dB HL at 0.5, 1, 2 and 4 kHz.
  Interventions: Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode

INTERVENTIONS:
Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode — During surgery using a retro-sigmoid approach in the cerebellopontine angle (microvascular decompression), near-field recording of human auditory nerve activity using a contact electrode is performed on patients with normal or impaired hearing threshold.
  Each patient is explored preoperatively by hearing tests. During the surgery, stimuli are delivered.

SUMMARY:
In humans, surface electrophysiological recordings of the cochlear nerve in response to a sound stimulus provide information about the cochlear's ability to encode sound. Depending on the stimulus, the fine structure and temporal envelope of the signal will vary, allowing us to determine its characteristics. By phenotyping patients before surgery using subjective and objective audiometric tests, it will be possible to isolate for each patient the moment when the fine structure disappears and when the temporal envelope is effective.

DETAILED DESCRIPTION:
During functional cerebellopontine angle surgery, a spherical electrode is placed on the human cochlear nerve to monitor hearing. Once the electrode is in place, clicks and speech signals with and without noise are delivered to analyze the cochlear electrophysiological signal produced. Depending on the characteristics recorded, this signal can be used to determine how fine structure and temporal envelope are encoded by the cochlea. Prior to surgery, each patient is evaluated by an audiologist to determine quiet and noise thresholds, tone and speech, electrocochleography, distortion testing, tympanometry, ABR and psychoacoustic testing.

ELIGIBILITY:
Inclusion criteria:

* The following will be included as hearing-impaired patients:

  * Male or female
  * Over 18 and up to 80 years of age
  * Normal otoscopic examination
  * Scheduled for surgery on the cerebellopontine angle (microvascular decompression)
  * With sensorineural hearing loss defined by average hearing thresholds between 21 dB HL and 40 dB HL at 0.5, 1, 2 and 4 kHz
  * Affiliated to a social security scheme
  * Having read the information note describing the study and having agreed in writing to participate by signing the informed consent form
* Will be included as normal-hearing patients:

  * Male or female
  * Over 18 and up to 80 years of age
  * Normal otoscopic examination
  * Scheduled for surgery on the cerebellopontine angle (microvascular decompression)
  * Free of sensorineural hearing loss, defined by average hearing thresholds of less than or equal to 20 dB HL in tonal air conduction audiometry, bilaterally on the side of the ear undergoing surgery and on the side not undergoing surgery, at 0.5, 1, 2 and 4 kHz
  * Affiliated to a social security scheme
  * Having read the information note describing the study and having agreed in writing to participate by signing the informed consent form

Exclusion criteria: patients will be excluded from the study if the auditory nerve is not accessible during surgery:

* Notably because of complete tumor invasion of the cochlear nerve (stage III and IV neuroma, advanced meningioma) ;
* Or because of a particular anatomical feature not identified during the preoperative examination, making its exposure for recordings impossible (protrusion of the posterior face of the rock).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To compare the amplitude of coding of complex and ecological sounds | At 48 months
  The goal is to compare the amplitude of coding of complex and ecological sounds (logatomes in the form of vowels or syllables: association of a consonant and a vowel) in the human auditory nerve between patients defined as normo and poorly hearing according to preoperative audiometric tests.
To compare the spectrum of coding of complex and ecological sounds | At 48 months
  The goal is to compare the spectrum of coding of complex and ecological sounds (logatomes in the form of vowels or syllables: association of a consonant and a vowel) in the human auditory nerve between patients defined as normo and poorly hearing according to preoperative audiometric tests.

SECONDARY OUTCOMES:
The spectrum of the temporal envelope of the signal | At 48 months
  To study the spectrum of the temporal envelope of the signal collected for each logatome in the general population studied and within the normal-hearing and hard-of-hearing groups.
The amplitude of the temporal envelope of the | at 48 months
  To study the amplitude of the temporal envelope of the signal collected for each logatome in the general population studied and within the normal-hearing and hard-of-hearing groups.
The spectrum of the fine structure of the signal | at 48 months
  To study the spectrum of the fine structure of the signal collected for each logatome in the general population studied and within the normal-hearing and hard-of-hearing groups.
The amplitude of the fine structure of the signal | at 48 months
  To study the amplitude of the fine structure of the signal collected for each logatome in the general population studied and within the normal-hearing and hard-of-hearing groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France